CLINICAL TRIAL: NCT03877679
Title: The Effect of Topical Curcumin Versus Topical Corticosteroid on Pain, Clinical Parameters and Salivary Level of IL-33 in Oral Lichen Planus Patients: A Randomized Controlled Clinical Trial
Brief Title: The Effect of Topical Curcumin Versus Topical Corticosteroid on Management of Oral Lichen Planus Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed salah abd-elhameed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMED2:5:1
Record Dates: First submitted 2018-09-24; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus; curcumin; IL-33; corticosteroids
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Triamcinolone; Orabase; Curcumin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor (CS) and statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- turmeric paste (Experimental): Topical curcumin gel (a mixture of curcumin powder and vegetable glycerin base in a ratio of 1:8 by weight) Mix with 85ml carbapol gel (125ml H2O + 0.5g carbapol + triethanolamine 3 drops) prepared in the Faculty of pharmacy-Cairo University traumeric extracted from Curcuma plant, it has anti-inflammatory, antioxidative and antineoplastic properties ((Nosratzehi et al., 2018), The curcumin is safe even in high doses, Since oxidative stress may play a role in pathophysiology of OLP, and by noting that OLP is a chronic inflammatory disease, the herbs which have both anti-inflammatory and antioxidant properties may efficiently control OLP (Kia et al., 2015).
  Interventions: Drug: Turmeric paste
- Triamcenolone in orabase (Active Comparator): Triamcenolone + na ploycarboxylate
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Triamcinolone — Triamcenolone +napolycarboxylate
  Other Names: Triamcenolone in orabase
  Arms: Triamcenolone in orabase
Drug: Turmeric paste — Topical turmeric paste (a mixture of curcumin powder and vegetable glycerin base in a ratio of 1:8 by weight) Mix with 85ml carbapol gel (125ml H2O + 0.5g carbapol + triethanolamine 3 drops) prepared in the Faculty of pharmacy-Cairo University
  Other Names: Curcumin
  Arms: turmeric paste

SUMMARY:
Introduce a new anti-inflammatory and antioxidant paste preparation (curcumin paste) in the management of Oral lichen planus.

* Assess the efficacy of this preparation on pain, clinical parameter and the level of IL-33 in saliva.
* Compare the outcome of new preparation with the gold standard treatment (corticosteroids).

DETAILED DESCRIPTION:
Two groups will be prepared then decision of which one take curcumin paste will be selected according to randomized numbers in a sequentially numbered, opaque, sealed envelope

1 group will take topical corticosteroid and 1 will take curcumin paste then IL-33 level in saliva will be measured at the base line and at the end of 4th week pain and clinical parameters will be measured at 2nd and 4th week

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be clinically diagnosed as having atrophic &/or erosive oral lichen planus.
* Patients with controlled diabetes and/or controlled hypertension will be included in the study.
* Patients with no history of taking corticosteroids for the last 6 months
* Patients who agrees to take medication.

Exclusion Criteria:

* Pregnant and lactating ladies.
* Patients with history of topical steroids during last 2 months & systemic steroids during last 6 months.
* Patients with recent dental filling associated with the lesion or associated with recent drug administration.
* Patient with uncontrolled diabetes, uncontrolled hypertension, or those with positive HCV ab or HBs Ag.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  measured by Visual Analog Scale (VAS) 0 = no pain 10= severe pain 0= no pain 10= pain severe pain

SECONDARY OUTCOMES:
clinical sign score | Baseline , 2nd week and 4th week
  measured by Thongprasom from score 0 to 5 0= only white lesion 5=area of erosion more than 2 cm
IL-33 level in saliva | base line and 4th week
  by ELISA

IPD SHARING:
Plan to Share IPD: Yes
All authors of this trial will have access to the final trial dataset.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after study completion
Access Criteria: pubmed

REFERENCES:
- [Background] Chainani-Wu N. Safety and anti-inflammatory activity of curcumin: a component of tumeric (Curcuma longa). J Altern Complement Med. 2003 Feb;9(1):161-8. doi: 10.1089/107555303321223035. PMID 12676044
- [Background] Greenberg G, Glick M. Burket's Oral Medicine: Diagnosis and Treatment. Hamilton, Ontario, BC Decker, 11th ed., 2008:90-1
- [Background] Nosratzehi T, Arbabi-Kalati F, Hamishehkar H, Bagheri S. Comparison of the Effects of Curcumin Mucoadhesive Paste and Local Corticosteroid on the Treatment of Erosive Oral Lichen Planus Lesions. J Natl Med Assoc. 2018 Feb;110(1):92-97. doi: 10.1016/j.jnma.2017.01.011. Epub 2017 May 11. PMID 29510851
- [Result] Chainani-Wu N, Silverman S Jr, Reingold A, Bostrom A, Mc Culloch C, Lozada-Nur F, Weintraub J. A randomized, placebo-controlled, double-blind clinical trial of curcuminoids in oral lichen planus. Phytomedicine. 2007 Aug;14(7-8):437-46. doi: 10.1016/j.phymed.2007.05.003. Epub 2007 Jul 2. PMID 17604143